CLINICAL TRIAL: NCT05433597
Title: A Two-blinded, Multicentre, Phase II/III RCT of Concurrent Chemo-radiotherapy Combined or Not Combined With TNF as the Therapy for Local-advancedNPC
Brief Title: A Two-blinded, Multicentre, Phase II/III RCT of Concurrent Chemo-radiotherapy Combined or Not Combined With TNF as the Therapy for LA-NPC
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Shanghai Weike Bioscience Co., Ltd. (Unknown)
Responsible Party: Principal Investigator, Yun-fei Xia, Principal Investigator, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2021-FXY-422
Record Dates: First submitted 2022-06-22; First posted 2022-06-27 (Actual); Last update posted 2022-06-27 (Actual); Status verified 2022-06

CONDITIONS: Nasopharyngeal Carcinoma; TNF; Chemo-radiotherapy
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Fluorouracil; Cisplatin; Radiotherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator): Chemotherapy: 5-fu: 200mg/m2/d, continuous intravenous infusion on the 1st to 30th day of each cycle; Cisplatin: 80mg/m2, used on the 1st and 28th day of each cycle; Q60d; Every 2 months for a treatment cycle, use 2 cycles, a total of 4 months.
  Radiotherapy: Radiotherapy was initiated on day 15 of the first cycle of chemotherapy GTV: 6810cGy (227 cGy/30f) Or 6996 cGy (212 cGy/ 33F); CTV: 5400-6000 cGy (180-200 cGy/f); Radiotherapy once a day, 5 times a week, a total of 30-33 times, a total of about 6 weeks.
  Placebo: Normal saline 1-2ml, intramuscular injection, QD, 30 days in the first and third months, once a day.
  Interventions: Drug: 5-fu; Drug: Cisplatin; Radiation: Radiotherapy; Drug: Placebo
- Experimental group (Active Comparator): Chemotherapy: 5-fu: 200mg/m2/d, continuous intravenous infusion on the 1st to 30th day of each cycle; Cisplatin: 80mg/m2, used on the 1st and 28th day of each cycle; Q60d; Every 2 months for a treatment cycle, use 2 cycles, a total of 4 months.
  Radiotherapy: Radiotherapy was initiated on day 15 of the first cycle of chemotherapy GTV: 6810cGy (227 cGy/30f) Or 6996 cGy (212 cGy/ 33F); CTV: 5400-6000 cGy (180-200 cGy/f); Radiotherapy once a day, 5 times a week, a total of 30-33 times, a total of about 6 weeks.
  Tianenfu (recombinant human tumor necrosis factor for injection) : 1 million IU (BSA<2.0m2) or 1.5 million IU (BSA≥2.0m2), dissolved in normal saline 1-2mL, intrascularization, QD, 30 days in the first and third months, once a day.
  Interventions: Drug: 5-fu; Drug: Cisplatin; Radiation: Radiotherapy; Drug: TNF

INTERVENTIONS:
Drug: 5-fu — 5-fu: 200mg/m2/d, continuous intravenous infusion on the 1st to 30th day of each cycle.
Drug: Cisplatin — Cisplatin: 80mg/m2, used on the 1st and 28th day of each cycle.
Radiation: Radiotherapy — Radiotherapy: Radiotherapy was initiated on day 15 of the first cycle of chemotherapy . GTV: 6810cGy (227 cGy/30f) Or 6996 cGy (212 cGy/ 33F); CTV: 5400-6000 cGy (180-200 cGy/f); Radiotherapy once a day, 5 times a week, a total of 30-33 times, a total of about 6 weeks.
Drug: TNF — TNF (recombinant human tumor necrosis factor for injection) : 1 million IU (BSA<2.0m2) or 1.5 million IU (BSA≥2.0m2), dissolved in normal saline 1-2mL, intramuscular, QD, 30 days in the first and third months, once a day.
  Arms: Experimental group
Drug: Placebo — Placebo: 1-2ml normal saline, intramuscular injection, QD, once a day, 30 days in the first and third months.
  Arms: Control group

SUMMARY:
Based on the application prospect of rmh-TNF combined with chemotherapy in the treatment of solid tumors. In this study, cisplatin combined with low dose 5-FU was proposed to enhance the immune function of 5-FU. Tianenfu is a novel recombinant modified human tumor necrosis with high activity and low toxicity. The fact that RMH-TNF has the potential of better in vivo efficacy and clinical antitumor effect. Therefore, the study was designed to investigate the treatment of concurrent chemoradiotherapy combined with TNF versus concurrent chemoradiotherapy combined with placebo for the efficacy and safety of advanced nasopharyngeal carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years old and ≤60 years old;
2. Pathologically confirmed nasopharyngeal carcinoma;
3. Patients with primary locally advanced non-metastatic nasopharyngeal carcinoma who were eligible for standard concurrent radiotherapy and chemotherapy were in line with stage III and IVA defined by the International Union against Cancer and American Joint Commission on Cancer (UICC/AJCC) staging System (version 8) (note: Stage III only included EBV-DNA>1×10^4 copy/mL).
4. Patients with locally advanced nasopharyngeal carcinoma who have not received prior radiotherapy or chemotherapy for the disease in this study;
5. Karnofsky functional status score should be at least 70 points (the decline of functional status score caused by tumor should be appropriately relaxed after the judgment of the researcher, and the minimum score should be no less than 50 points. );
6. At least 1 measurable lesion according to RECIST1.1 assessment criteria, measurable lesion should not have received local treatment such as radiotherapy;
7. Expected survival ≥3 months;
8. The function of vital organs meets the following requirements (not allowed within 14 days before screening . May use any blood components, cell growth factors, leukoplast, platelets Drugs, anemia correction drugs) :

   * Neutrophil absolute count (ANC) ≥1.5×109/L
   * Platelet ≥100×109/L;
   * Hemoglobin ≥8.0g/ dL (note: Hemoglobin ≥8.0g/ dL can be achieved through blood transfusion or other intervention);
   * Serum albumin ≥2.8g/dL;
   * Bilirubin ≤ 1.5x ULN, ALT and AST≤ 1.5x ULN; ALT and AST≤ 5x ULN if liver metastasis was present;
   * creatinine clearance ≥50mL/min
9. Women of non-surgical sterilization or reproductive age and sexually active men enrolled in the study are required to use a medically effective form of contraception (such as an intrauterine device [IUD], birth control pills or condoms) for the duration of the study treatment and for at least 3 months after the last use of Tamfu and for at least 6 months after the last use of chemotherapy; The serum or urine HCG test of female patients of reproductive age who were not undergoing surgical sterilization must be negative within 7 days prior to study enrollment. And must be non lactation period; 10 Informed consent has been signed. -

Exclusion Criteria:

1. Have a history of allergy to 5-FU, cisplatin and tumor necrosis factor;
2. Previous treatment related to tumor necrosis factor (TNF);
3. Major surgery other than nasopharyngeal cancer was diagnosed within 28 days prior to randomization or major surgery was expected during the study period;
4. The subject has any active autoimmune disease or a history of autoimmune disease (e.g., but not limited to: interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism); Subjects with vitiligo or asthma in complete remission during childhood without any intervention as adults could be included; Subjects with asthma requiring medical intervention with bronchodilators were excluded);
5. Subject is taking immunosuppressants, or systemic, or absorbable sites Hormone therapy to achieve immunosuppression (dose >10mg/ day prednisone or Other equally effective hormones) and continued to be used within 2 weeks prior to enrollment.
6. The subject has previous or co-existing malignancies (except those that have been cured and survived for more than 5 years without cancer, such as basal cell carcinoma of the skin, carcinoma in situ of the cervix and papillary carcinoma of the thyroid);
7. Patients with cardiac clinical symptoms or diseases that are not well controlled, such as: ① HEART failure of NYHA grade 2 or above ② unstable angina pectoris ③ myocardial infarction within 1 year ⑤ clinically significant ventricular arrhythmias or ventricular arrhythmias requiring treatment or intervention;
8. Subjects have active infection or have unexplained fever >38.5 degrees during screening but before the first dose (the investigator judged that the subjects' fever due to tumor could be included in the study);
9. Subjects with congenital or acquired immune deficiency (e.g. HIV infected), or active hepatitis (reference: HBsAg, anti-HBS, HBeAg, anti-HBC, anti-HBE, HBV DNA≥10⁴/ml, liver cell transaminase, etc.); Hepatitis C reference: HCV antibodies and HCVRNA);
10. The subject has a known history of psychotropic drug abuse, alcoholism or drug abuse;
11. In the judgment of the researcher, the subject has other factors that may lead to the termination of the study, such as other serious diseases (including mental diseases) requiring combined treatment, serious abnormal laboratory examination, family or social factors, which may affect the safety of the subject, or the collection of test data and samples.
12. Women who are pregnant or breastfeeding, or who refuse/cannot accept medically acceptable conditions. For women with potential pregnancy and sexually active men.

    -

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 172 (Estimated)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2024-07-01 (Estimated); Study Completion 2029-07-01 (Estimated)

PRIMARY OUTCOMES:
OS | Up to 5 years
  Overall survival Overall survival Overall survival Overall survival Overall survival Overall survival Overall survival Overall survival
PFS | Up to 5 years
  Progression-free survival
Severe drug-related adverse events | Up to 2 approximately years
  grade III-V according to CTCAE v4.0

SECONDARY OUTCOMES:
ORR | Up to 2 approximately years
  Objective response rate
DCR | Up to 2 approximately years
  Disease control rate
DOR | Up to 2 approximately years
  Duration of response
Drug-related adverse events grade I-II | Up to 2 approximately years
  Minor drug-related adverse events grade I-II according to CTCAE v4.0

CONTACTS AND LOCATIONS:
Overall Officials: Yun-fei Xia, MD, Principal Investigator — Sun Yat-sen University

IPD SHARING:
Plan to Share IPD: No